CLINICAL TRIAL: NCT05147727
Title: A Single-center, Open-label, Fixed-sequence Study to Evaluate the Effects of Fluconazole on the Pharmacokinetics and Safety of Famitinib in Healthy Subjects
Brief Title: Drug-drug Interaction Study Between Fluconazole and Famitinib in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FMTN-I-108
Record Dates: First submitted 2021-12-06; First posted 2021-12-07 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Fluconazole and famitinib interaction
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluconazole and Famitinib interaction (Experimental)
  Interventions: Drug: Fluconazole、Famitinib

INTERVENTIONS:
Drug: Fluconazole、Famitinib — Fluconazole, once daily on Days 12 to 24; Famitinib, once daily on Days 1 and 15

SUMMARY:
An open-label, fixed-sequence, drug-drug interaction study to evaluate the effects of fluconazole on the pharmacokinetics and safety of famitinib in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. With my consent and informed consent, I am willing and able to complete the study in accordance with the requirements of the experimental protocol;
2. Healthy male or female aged 18-45 years (including threshold) on the date of signing the informed consent form;
3. Male body weight ≥ 50 kg, female body weight ≥ 45 kg, body mass index (BMI) in the range of 19.0-26.0 kg / m2 (including the critical value);
4. Physical examination, vital signs, laboratory measurements (blood routine, blood biochemistry, urine routine test, coagulation function, etc.), 12-lead ECG, abdominal B-ultrasound, chest X-ray, etc. are normal or abnormal, but the researcher has no clinical significance according to NCI CTCAE 5.0 standard;
5. Fertile subjects had no family planning and had to take acceptable contraceptive measures and no plans to donate eggs and sperm within 3 months from the date of signing informed consent to the last medication; the serum pregnancy test of fertile women within 24 hours before the first administration of the study drug should be negative.

Exclusion Criteria:

1. Those who have previously suffered from primary diseases of important organs, including but not limited to neuropsychiatric, cardiovascular, digestive tract, respiratory system, urinary, endocrine, blood, immune and other diseases, which are judged by the researchers to be unsuitable for the trial;
2. Subjects who have received any previous operation affecting gastrointestinal absorption;
3. Subjects who had received any surgery within 6 months before screening, or planned to undergo surgery during the study period;
4. Those who lost blood or donated more than 400 ml or received blood transfusion within 3 months before screening;
5. HBsAg positive, HCVAb positive, HIV antibody positive, syphilis antibody positive;
6. History of drug use in the past 5 years or drug abuse, or drug screening positive;
7. Smoking and alcohol addict and unable to stop smoking during the test period; those with positive alcohol screening; those with positive nicotine screening;
8. Subjects who have swallowing resistance or obstacle that will affect the drug absorption;
9. Allergic constitution, including severe drug allergy or drug allergy history; known allergy to fluconazole and famitinib or its excipients;
10. Those who have participated in other clinical trials and taken the study drug within 3 months before taking the study drug for the first time;
11. Inducers or inhibitors of CYP3A4 were taken within 4 weeks before the first administration of study drug;
12. Taking any prescription drug, over-the-counter drug, traditional Chinese medicine or food supplement within 2 weeks before taking the study drug for the first time;
13. Ingestion of grapefruit containing products, fruit juice, food or beverage containing methylxanthine or alcohol within 48 hours before taking the study drug for the first time; taking strenuous exercise; or having other factors affecting the absorption, distribution, metabolism and excretion of drugs;
14. Lactating women;
15. The researchers considered that the subjects had any other factors that were not suitable for the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Maximum observed serum concentration (Cmax) for famitinib | Day 1 to Day 25
Area under the concentration-time curve from time zero to time t (AUC0-t,) for famitinib | Day 1 to Day 25
Area under the concentration-time curve extrapolated to infinity (AUC0-∞.) for famitinib (if applicable) | Day 1 to Day 25

SECONDARY OUTCOMES:
Time to maximum observed serum concentration (Tmax) for famitinib | Day 1 to Day 25
Time to elimination half-life (t1/2) for famitinib | Day 1 to Day 25
Apparent oral clearance (CL/F) for famitinib | Day 1 to Day 25
Apparent Volume of Distribution (Vz/F) for famitinib | Day 1 to Day 25
Tmax for famitinib metabolite SHR116637 | Day 1 to Day 25
Cmax for famitinib metabolite SHR116637 | Day 1 to Day 25
AUC0-t, for famitinib metabolite SHR116637 | Day 1 to Day 25
AUC0-∞. for famitinib metabolite SHR116637(if applicable) | Day 1 to Day 25
t1/2 for famitinib metabolite SHR116637 | Day 1 to Day 25
The incidence and severity of adverse events/serious adverse events (based on NCI-CTC AE 5.0) | Day 1 to Day 25

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided